CLINICAL TRIAL: NCT06136338
Title: Effectiveness of Mindfulness Intervention to Determine the Timing of Labor Admission, Uncertainty and Anxiety Among Pregnant Women: A Pilot Study.
Brief Title: A Pilot Study of Mindfulness Intervention to the Timing of Labor Admission, Uncertainty and Anxiety
Acronym: MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chia-Wen Lee, assistant professor, National Taipei University of Nursing and Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: C109037
Record Dates: First submitted 2023-11-08; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Anxiety; Uncertain Viability of Pregnancy
Keywords: mindfulness-based intervention; childbirth related anxiety; childbirth related uncertainty
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Experimental group： intervention + routine care Control group：routine care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness intervention group (Experimental): intervention + routine care
  Interventions: Behavioral: Mindfulness training
- Control group (No Intervention): routine care

INTERVENTIONS:
Behavioral: Mindfulness training — Women in the experimental group underwent four sessions of mindfulness training. The mindfulness training started at the 28th week of pregnancy for the women, the second training was at the 30th week of pregnancy, the third was at the 32nd week of pregnancy, and the last was at the 34th week of pregnancy, with each session lasting 45 minutes.
  Arms: Mindfulness intervention group

SUMMARY:
The goal of this quasi-experienmental study is to investigate the effectiveness of mindfulness-based intervention in the level of uncertainty and anxiety, and determintation towards hospital admission among pregnant women. The main questions : • Do pregnant women in intervention group reduce anxiety and uncertainty? • Do pregnant women in intervention group increase self-determintation ability towards hospital admission? Women in the intervention group participated 4 weeks mindfulness-based intervention online courses, Researchers have seen effectiveness of mindfulness-based intervention in the level of uncertainty, anxiety, and determintation towards hospital admission among pregnant women.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effectiness of mindfulness-based intervention in the level of uncertainty and anxiety, and determination towards hospital admission among pregnant women. This study is a quasi-experimental design and convenient sampling to recruit primipara women in the distrct hospital. A total of 31 participants were enrolled, eleven participatns were assigned to the experimental group, and twenty participants were in the control group. The measurements were demographic characteristics andobstetric data, FFMQ,VAS of uncertainty and anxiety, and ACS.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years old.
2. Single primiparous women with gestation over 28 weeks.
3. Clear consciousness, ability to speak, write and read Chinese, able to write questionnaires by themselves.
4. Those who are expected to have a vaginal delivery.
5. Agree to participate in the researcher after the research description.

Exclusion Criteria:

1. People with mental health problems, such as: depression, mental illness, etc.
2. The woman has pregnancy complications or the fetus has any complications.
3. Arrange for labor induction.
4. Those who have meditated or attended mindfulness courses.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-03-23 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
measure of dispositional mindfulness on the Five Facets Mindfulness Questionnaire（FFMQ） | 28th week gestational, 34th gestational week and 3-days postpartum
  The Five Facet Mindfulness Questionnaire(FFMQ) is a 39-item self-report measure of dispositional mindfulness. The scale is comprised of five factors: Observing, describing, acting with awareness, nonjudging, and nonreacting. The FFMQ has demonstrated strong psychometric properties.Each item is rated on a five-point Likert-type scale ranging from never or very rarely true to very often or always true. The total score range from 39-195, higher scores mean a better outcome.
Uncertainty Visual Analogue Scale to measure the degree of uncertainty of women about admission to the hospital | 28th week gestational, 34th gestational week and 3-days postpartum
  This study uses a visual analog scale of 0-10 points, the score ranges from 0 to 10 points, the higher score, means the women is more sense of uncertainty.
Anxiety Visual Analogue Scale to measure the women overall anxiety | 28th week gestational, 34th gestational week and 3-days postpartum
  This study uses a visual analog scale of 0-10 points, the score ranges from 0 to 10 points, the higher score, means the women is more anxiety.
If women improve attention will help them to make decision, so measure of decision making ability on Attentional Control Scale(ACS) | 28th week gestational, 34th gestational week and 3-days postpartum
  The Attentional Control Scale (ACS) measures the ability to focus attention, to shift attention between tasks, and to flexibly control one's thoughts.This 20-item, self-report questionnaire examines one's ability to control one's attention.Participants answered questions based on a four-point scale ranging from almost never to always. The total score range from 20-80, higher scores mean a better outcome.
labor and childbirth information | 3-days postpartum
  This part of the information is transcribed from the medical records. Data include: who decides to be admitted to the hospital, how many time was admissions rejections, the situation of the first vaginal examination when admitted to the hospital, and the uterus contraction pressure and frequency, duration of labor, labor-inducing drugs, epidural pain relief usage, delivery method, assisted delivery.

CONTACTS AND LOCATIONS:
Overall Officials: LEE Chia-Wen, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No